CLINICAL TRIAL: NCT05442567
Title: A Phase 3b Extension Study to Evaluate the Long-term Safety of Vedolizumab Intravenous in Pediatric Patients With Ulcerative Colitis or Crohn's Disease
Brief Title: A Study of Vedolizumab in Children With Ulcerative Colitis (UC) or Crohn's Disease (CD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN0002-3029; 2023-509046-36-00 (EU CTIS Number: EU CT Number); jRCT2071230036 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-06-30; First posted 2022-07-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Treatment Cohort: Participants 10 to ≤15 kg, Vedolizumab 150 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing 10 to ≤15 kg will receive vedolizumab 150 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Treatment Cohort: Participants 10 to ≤15 kg, Vedolizumab 100 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing 10 to ≤15 kg will receive vedolizumab 100 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Treatment Cohort: Participants >15 to <30 kg, Vedolizumab 200 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing >15 to <30 kg will receive vedolizumab 200 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Treatment Cohort: Participants >15 to <30 kg, Vedolizumab 100 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing >15 to <30 kg will receive vedolizumab 100 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Treatment Cohort: Participants ≥30 kg, Vedolizumab 300 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing ≥30 kg will receive vedolizumab 300 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Treatment Cohort: Participants ≥30 kg, Vedolizumab 150 mg (Experimental): Eligible participants from studies MLN0002-3024 or MLN0002-3025 weighing ≥30 kg will receive vedolizumab 150 mg, IV infusion, Q8W, (same as their Week 46 dose in parent study) in this study for up to approximately 5 years.
  Interventions: Drug: Vedolizumab IV
- Observational Cohort: Early Terminated Participants From Parent Studies (Other): Participants will have assessment visits at Day 1 and Weeks 8, 34, 60, and 86 as part of a long-term follow-up period to assess prespecified safety events of interest and to monitor growth and pubertal development for approximately 2 years after their last dose of study drug in parent study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Other Names: MLN0002; ENTYVIO; KYNTELES
  Arms: Treatment Cohort: Participants 10 to ≤15 kg, Vedolizumab 100 mg; Treatment Cohort: Participants 10 to ≤15 kg, Vedolizumab 150 mg; Treatment Cohort: Participants >15 to <30 kg, Vedolizumab 100 mg; Treatment Cohort: Participants >15 to <30 kg, Vedolizumab 200 mg; Treatment Cohort: Participants ≥30 kg, Vedolizumab 150 mg; Treatment Cohort: Participants ≥30 kg, Vedolizumab 300 mg
Other: No Intervention — Participants will not receive any intervention in the Observational Cohort.
  Arms: Observational Cohort: Early Terminated Participants From Parent Studies

SUMMARY:
The study is an extension of two parent studies (MLN0002-3024 [NCT04779307] and MLN0002-3025 [NCT04779320]). Participants must have participated in one of the previous studies. The purpose of this study is to collect the long-term safety of vedolizumab in children with UC or CD.

DETAILED DESCRIPTION:
This multi-center trial is conducted worldwide. Up to 240 patients would be enrolled from Studies MLN0002-3024 [participants with UC] and MLN0002-3025 [participants with CD], either in the Treatment Cohort or in the Observational Cohort. Approximately 93 participants who have previously participated either in study MLN0002-3024 or MLN0002-3025, referred to as parent study, are expected to roll over to the MLN0002-3029 study in the treatment cohort.

Treatment Cohort:

The drug being tested in this study is called vedolizumab, being studied to treat pediatric patients who have UC or CD.

Participants eligible for the Treatment Cohort can be administered vedolizumab intravenous (IV) at Week 54 visit of parent study or up to 1 week after Week 54 of the parent study based on the availability of test results needed to assess eligibility of the participant. At this study entry, participants will be administered the same blinded dose of vedolizumab IV that was received at Week 46 in the parent study and will then continue to receive vedolizumab IV at a frequency of once every 8 weeks (Q8W) in the following treatment groups:

* Participants 10 to ≤15 kilogram (kg), Vedolizumab 150 milligram (mg) (High dose)
* Participants 10 to ≤15 kg, Vedolizumab 100 mg (Low dose)
* Participants >15 to <30 kg, Vedolizumab 200 mg (High dose)
* Participants >15 to <30 kg, Vedolizumab 100 mg (Low dose)
* Participants ≥30 kg, Vedolizumab 300 mg (High dose)
* Participants ≥30 kg, Vedolizumab 150 mg (Low dose)

Blinding of dose group assignment of the parent study will continue until the respective parent study is unblinded in order to protect the blinding of the parent study.

The overall time to participate in the Treatment Cohort of this study is up to participant withdrawal, or until vedolizumab IV is commercially available for pediatric indication(s) in the participant's country or until other drug access programs become available, or Sponsor's decision for study closure, or for up to approximately 5 years, whichever comes first. Participants who complete or are discontinued from the study for any reason will complete the final safety/end of study (EOS) visit 18 weeks after their last dose of study drug.

Observational Cohort:

Participants who received at least 1 dose of study drug during parent study and early terminated or are not eligible for the Treatment Cohort of this study after completion of the Week 54 visit of parent study, will be enrolled in the Observational Cohort of this study as part of a long-term follow-up period to assess prespecified safety events of interest and will not receive continued treatment with vedolizumab IV.

The overall time to participate in the Observational Cohort is up to approximately 2 years.

ELIGIBILITY:
Main Inclusion Criteria:

For Treatment Cohort:

1. The participant should have completed Study MLN0002-3024 or Study MLN0002-3025 and achieved corticosteroid-free clinical response at Week 54 (and has tapered off of steroids, as applicable, at least 12 weeks before Week 54) as defined by a reduction of partial Mayo score of ≥2 points and ≥25% from baseline for participants with UC, or by a decrease of pediatric Crohn's disease activity index (PCDAI) of ≥15 points for participants with CD and with total PCDAI ≤30.
2. A male participant who is sexually active with a female partner of childbearing potential agrees to use a barrier method of contraception (e.g., condom with or without spermicide) from signing of participant/parental informed consent and/or pediatric assent throughout the duration of the study and for 18 weeks after last dose. The female partner of a male participant should also be advised to use a highly effective method of contraception.
3. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use a highly effective method of contraception from signing of participant/parental informed consent and/or pediatric assent throughout the duration of the study and 18 weeks after the last dose.

For Observational Cohort:

1. The participant has received at least 1 dose of vedolizumab during Study MLN0002-3024 or Study MLN0002-3025 and early terminated OR completed the Week 54 visit of Study MLN0002-3024 or Study MLN0002-3025 but was not eligible to enroll in the treatment cohort of this study.

Main Exclusion Criteria:

For Treatment Cohort only:

1. The participant currently requires major surgical intervention for UC or CD (e.g., bowel resection), or is anticipated to require major surgical intervention for UC or CD during the study.
2. The participant has developed any new unstable or uncontrolled cardiovascular, heart failure moderate to severe (New York Class Association III or IV), pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, coagulation, immunological, endocrine/metabolic, neurological, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
3. The participant has other serious comorbidities that will limit their ability to complete the study.
4. The participant is unable to comply with all study assessments.
5. The participant has hypersensitivity or allergies to any of the vedolizumab excipients.
6. The participant is lactating or pregnant.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2031-08-15 (Estimated); Study Completion 2031-08-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Cohort: Number of Participants With at Least One Adverse Event (AE) | From first dose of study drug up to approximately 5 years
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have causal relationship with this treatment. AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether or not it is considered related to drug.
Observational Cohort: Number of Participants With Prespecified Safety Events | Up to approximately 2 years
  Prespecified safety events will include serious infections, malignancies, progressive multifocal leukoencephalopathy (PML), concerns about growth and pubertal development, and bowel surgery.

SECONDARY OUTCOMES:
Treatment Cohort: Time to Major Inflammatory Bowel Disease (IBD)-related Events | Up to approximately 5 years
  Major IBD-related events include hospitalizations, surgeries, and procedures in pediatric participants with UC or CD.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Total Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III questionnaire is a self-reported measure with 35 closed questions encompassing 6 domains: Bowel Symptoms (7 items), Systemic Symptoms (3 items), Social Functioning (12 items), Body Image (3 items), Treatment/Interventions (3 items), and Emotional Functioning (7 items). The IMPACT-III uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The total score is an average of all item scores. The outcome score ranges from 35 to 175, with higher scores suggesting better quality of life. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Bowel Symptom Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Bowel Symptom Subscale is a self-reported measure with 7 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The bowel symptom subscale score ranges from 1 to 35, with higher scores indicating lesser bowel symptoms. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Systemic Symptom Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Systemic Symptom Subscale is a self-reported measure with 3 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The Systemic symptom subscale score ranges from 1 to 15, with higher scores indicating lesser systemic symptoms. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Social Functioning Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Social Functioning Subscale is a self-reported measure with 12 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The social functioning subscale score ranges from 1 to 60, with higher scores indicating better social functioning. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Body Image Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Body Image Subscale is a self-reported measure with 3 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The body image subscale score ranges from 1 to 15, with higher scores indicating better body image. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Treatment/Intervention Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Treatment/Intervention Subscale is a self-reported measure with 3 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The treatment/intervention subscale score ranges from 1 to 15, with higher scores indicating ease of administration of treatment/interventions. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.
Treatment Cohort: Change From Baseline of Studies MLN0002-3024 (UC) or MLN0002-3025 (CD) in IMPACT-III Emotional Functioning Subscale Score for Participants Aged 9 to 17 Years for Every 24 Weeks | Baseline, every 24 weeks in this study (up to approximately 5 years)
  The IMPACT-III Emotional Functioning Subscale is a self-reported measure with 7 closed questions. It uses a 5-point Likert scale ranging from 1 (bad 'quality of life' condition) to 5 (good 'quality of life' condition) for all answers. The emotional functioning subscale score ranges from 1 to 35, with higher scores indicating better emotional functioning. This outcome will be assessed in participants who were aged 9 to 17 years at the time of first dose of study drug in study MLN0002-3024 or MLN0002-3025. Baseline refers to the Baseline of study MLN0002-3024 or MLN0002-3025.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (68):
- United States (14):
  - Phoenix Childrens Hospital -1919 E Thompson Rd, Phoenix, Arizona
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - Childrens Center For Digestive Healthcare, Atlanta, Georgia
  - Advocate Children's Hospital Park Ridge, Park Ridge, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - MNGI Digestive Health PA-Plymouth, Minneapolis, Minnesota
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Goryeb Children's Hospital, Morristown, New Jersey
  - The Steven and Alexandra Cohen Childrens Medical Center of New York - BRANY - PPDS, New Hyde Park, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Carilion Children's Tanglewood Center, Roanoke, Virginia
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Brussel - PIN, Jette, Brussels Capital
  - UZ Leuven, Leuven, Vlaams Brabant
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
- China (4):
  - Beijing Children Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Henan Children's Hospital (Zhengzhou Children's Hospital), Zhengzhou, Henan
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Children's Hospital Zhejiang UniversitySchool of Medicine, Hangzhou, Zhejiang
- Klinika Za Djecje Bolesti Zagreb, Zagreb, City of Zagreb, Croatia
- Greece (3):
  - Attikon University General Hospital, Athens, Attica
  - Children's Hospital "Agia Sofia", Athens
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc, Borsod-Abauj Zemplen county
  - Semmelweis Egyetem, Budapest
- Israel (6):
  - Schneider Childrens Medical Center of Israel Petah Tikvah PIN, Petah Tikva, Central District
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Rambam Medical Center - PPDS, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (6):
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda USL di Bologna, Bologna, Emilia-Romagna
  - Sapienza University of Rome, Rome, Lazio
  - Fondazione IRCCS San Gerardo dei Tintori - ASST di Monza A. O. San Gerardo, Monza, Lombardy
  - Universita degli Studi di Padova, Padua, Veneto
- Japan (4):
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - National Center for Child Health and Development, Setagaya-Ku, Tokyo
- Poland (8):
  - Uniwersytecki Szpital Dzieciecy, Krakow, Lesser Poland Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Masovian Voivodeship
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - Gornoslaskie Centrum Zdrowia Dziecka Im. Sw. Jana Pawla II Spsk Nr 6 Sum W Katowicach, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Narodny ustav detskych chorob, Bratislava, Slovakia
- South Korea (4):
  - Kyungpook National University Chilgok hospital, Daegu, Daegu Gwang'yeogsi
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul
- United Kingdom (5):
  - Great Ormond Street Hospital (GOSH), London, London, City of
  - Noahs Ark Childrens Hospital for Wales - PPDS - PIN, Cardiff, South Glamorgan
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Barts Health NHS Trust, London
  - Royal Manchester Children's Hospital - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/ef380ef1e1ac489a?idFilter=%5B%22MLN0002-3029%22%5D